CLINICAL TRIAL: NCT00001364
Title: Evaluation and Treatment of Patients With Spinal Vascular Abnormalities
Brief Title: Evaluation and Treatment of Patients Spinal Blood Vessel Abnormalities
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 930151; 93-N-0151
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-12-10

CONDITIONS: Arteriovenous Fistula; Arteriovenous Malformation; Spinal Cord Disease
Keywords: Spinal Arteriovenous Malformations; Spinal Dural Arteriovenous Fistulas; Surgery; Embolization; Spinal Arteriography
MeSH Terms: conditions — Arteriovenous Fistula; Arteriovenous Malformations; Spinal Cord Diseases

SUMMARY:
Arteriovenous malformations (AVM) are abnormally formed blood vessels that can be located throughout the brain and spinal cord. Patients with abnormalities of the blood vessels located in and around the spinal cord can develop many neurological problems. Some problems include, weakness, pain, difficulty walking, paralysis, and even death.

The treatment for these AVMs depends on their location, the type of malformation, the area of the spine involved, and the condition of the patient at the time of treatment. The treatment is aimed at stopping the neurologic problems from worsening and possibly correcting the existing problems. There are two commonly used treatments for AVMs, surgery and embolization (blocking off of blood flow to the AVM).

However, researchers have limited experience treating these conditions because they are rare. In addition, it has been difficult to classify different kinds of AVMs and to develop new treatments for them.

This study is designed to increase researchers understanding of AVMs by admitting and following patients diagnosed with the condition. By increasing the amount of patients studied diagnosed with spinal blood vessel abnormalities, researchers can begin to develop new management plans for patients with AVMs.

DETAILED DESCRIPTION:
Spinal Arteriovenous Malformations are rare lesions that frequently effect young patients and adults in their most productive years. They cause progressive myelopathy, ultimately causing paraplegia or quadriplegia if untreated. Because they are rare lesions, experience with treating them in sufficient numbers to permit classification of them, investigation of the pathophysiology of myelopathy, and the introduction of new techniques for treatment has been possible in only a very few centers in this country. One essential element of investigation of them is selective spinal arteriography. Since selective spinal arteriography was first introduced for these lesions here at the NIH in the mid 1960's by Drs. John Doppman and Giovanni DiChiro, the NIH has been such a center of expertise for patients with spinal arteriovenous malformations. Because of this, NIH has been, and is, a national referral center for these patients. However, there has never been an approved protocol at the NIH for investigation or treatment of these patients. The purpose of this proposal is to present a plan of investigation and treatment which will serve as a protocol under which to admit these patients and to permit continued accrual of clinical experience with them that will serve to guide others in the management of these patients.

ELIGIBILITY:
* INCLUSION CRITERIA:

Adult greater than or equal to 18 years with known or suspected spinal AVM and capacity to provide written informed consent.

Child ages 4-18 with known or suspected spinal AVM and with parent/guardian informed consent.

EXCLUSION CRITERIA:

Unable to tolerate MRI and/or spinal arteriography.

Child less than 4 years.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 1993-06-02; Study Completion 2007-12-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Oldfield EH, Doppman JL. Spinal arteriovenous malformations. Clin Neurosurg. 1988;34:161-83. No abstract available. PMID 3288393